CLINICAL TRIAL: NCT05716893
Title: Phase 2 Trial of Adaptive Versus Standard Dosing of Aerobic Training in Patients Receiving Chemotherapy for Primary Breast Cance
Brief Title: Study of Aerobic Training for People Receiving Chemotherapy for Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-364
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Breast Carcinoma
Keywords: Breast cancer; Breast carcinoma; Primary breast cancer; Aerobic Training; 22-364; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive Aerobic Training/AT Dosing (Experimental): Participants with newly diagnosed primary breast cancer initiating chemotherapy.
  Interventions: Behavioral: Adaptive Aerobic Training/AT Dosing
- Standard (fixed) Aerobic Training/AT dosing (Active Comparator): Participants with newly diagnosed primary breast cancer initiating chemotherapy.
  Interventions: Behavioral: Standard (fixed) Aerobic Training/AT dosing

INTERVENTIONS:
Behavioral: Adaptive Aerobic Training/AT Dosing — o In Phase A (~32 weeks), AT will consist of supervised walking delivered up to 7 days per week using an adaptive dosing schedule that starts at 90 min/wk and is escalated 30 min/wk every 2 weeks to a maximal dose of 300 mins/wk. In Phase B (~20 weeks), AT will consist of supervised adaptive AT dosing in patients with a CRF Δ<3.50 ml O2 .kg-1.min-1 from baseline to ~32 weeks, or unsupervised AT in patients with a CRF Δ>3.50 ml O2 .kg-1.min-1 from baseline to ~32 weeks. Supervised AT will be monitored using TeleEx.
  Arms: Adaptive Aerobic Training/AT Dosing
Behavioral: Standard (fixed) Aerobic Training/AT dosing — In Phase A (~32 weeks), AT will consist of supervised walking delivered up to 7 days per week to achieve a cumulative total duration of: 90 min/wk (standard fixed dosing). In Phase B (~20 weeks), AT will consist of supervised adaptive AT dosing in patients with a CRF Δ<3.50 ml O2 .kg-1.min-1 from baseline to ~32 weeks, or unsupervised AT in patients with a CRF Δ>3.50 ml O2 .kg-1.min-1 from baseline to ~32 weeks. Supervised AT will be monitored using TeleEx.
  Arms: Standard (fixed) Aerobic Training/AT dosing

SUMMARY:
In this study, investigators will compare standard Aerobic Training/AT with adaptive Aerobic Training/AT. Standard AT will be a fixed (unchanging) amount of walking each week, while adaptive AT will adjust the level of exercise depending on participants' response to the exercise. Investigators will see how both study approaches (standard AT and adaptive AT) affect participants' CRF.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Female
* Diagnosed with primary breast cancer as defined by one of the following:

  * Histological confirmation
  * As per standard of care imaging
* Scheduled to receive neoadjuvant/adjuvant chemotherapy
* Performing ≤90 minutes of moderate- and/or strenuous-intensity exercise per week, as evaluated by self-report
* Willingness to comply with all study-related procedures
* Able to achieve an acceptable peak baseline CPET, as defined by any of the following criteria:

  1. Achieving a plateau in oxygen consumption, concurrent with an increase in power output;
  2. A respiratory exchange ratio ≥ 1.10;
  3. Attainment of maximal predicted heart rate (HRmax) (i.e., within 10 bpm of age-predicted HRmax [HRmax = 220-Age[years]);
  4. Volitional exhaustion, as measured by a rating of perceived exertion (RPE) ≥ 18 on the BORG scale.

Exclusion Criteria:

* Enrollment onto any other interventional investigational study, except interventions determined by the PI not to confound study outcomes
* Receiving treatment for any other diagnosis of invasive cancer
* Distant metastatic malignancy of any kind
* Mental impairment leading to inability to cooperate
* Any of the following contraindications to cardiopulmonary exercise testing:

  i. Acute myocardial infarction within 3-5 days of any planned study procedures; ii. Unstable angina; iii. Uncontrolled arrhythmia causing symptoms or hemodynamic compromise; iv. Recurrent syncope; v. Active endocarditis; vi. Acute myocarditis or pericarditis; vii. Symptomatic severe aortic stenosis; viii. Uncontrolled heart failure; ix. Acute pulmonary embolus or pulmonary infarction within 3 months of any planned study procedures; x. Thrombosis of lower extremities; xi. Suspected dissecting aneurysm; xii. Uncontrolled asthma; xiii. Pulmonary edema; xiv. Respiratory failure; xv. Acute non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (i.e., infection, renal failure, thyrotoxicosis) xvi. Room air desaturation at rest ≤ 85%
* Any other condition or intercurrent illness that, in the opinion of the investigator, makes the subject a poor candidate for study participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness (CRF) response rate | 32 weeks from baseline
  The primary endpoint will be CRF response rate as assessed by the proportion of patients with a peak oxygen consumption (VO2peak; ml O2 .kg-1.min-1 ) change from baseline (T0) to T2 (~32 weeks) of ≥3.50 ml O2 .kg-1.min-1 . A CRF change ≥3.50 ml O2 .kg-1.min-1 will be considered a response; a change <3.50 ml O2 .kg-1.min-1 will be considered a non-response.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Scott, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org